CLINICAL TRIAL: NCT05988671
Title: Comparison of Intraperitoneal Dexamethasone, Dexmedetomidine, and Dexamethasone-Dexmedetomidine Combination on Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy: A Randomized Clinical Trial
Brief Title: Intraperitoneal Dexamethasone, Dexmedetomidine, and Dexamethasone-Dexmedetomidine Combination on Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC 10-3-2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Saline Solution; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): received 20 ml normal saline
  Interventions: Drug: normal Saline
- dexamethasone group (Active Comparator): received 8mg dexamethasone
  Interventions: Drug: Dexamethasone
- dexmedetomidine group (Active Comparator): received dexmedetomidine 1mic/kg
  Interventions: Drug: Dexmedetomidine
- combined group (Active Comparator): received combination of both 8mg dexamethasone+ dexmedetomidine 1mic/kg
  Interventions: Drug: Combination of dexamethasone + dexmedetomidine

INTERVENTIONS:
Drug: normal Saline — Intraperitoneal route
  Arms: Control group
Drug: Dexamethasone — Intraperitoneal route
  Arms: dexamethasone group
Drug: Dexmedetomidine — Intraperitoneal route
  Arms: dexmedetomidine group
Drug: Combination of dexamethasone + dexmedetomidine — Intraperitoneal route
  Arms: combined group

SUMMARY:
Nausea and vomiting are some of the most common complaints of patients after any anesthesia, which is often associated with postop-erative pain. The double-blind clinical trial study aimed to compare the prophylactic effect of dexamethasone and dexmedetomidine and their combination in reducing postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 - 50 years
* ASA I OR II
* undergo laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with history of psychotic illnesses,
* Parkinson's disease
* motion disorder
* Smoker
* or history of chemotherapy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The number of patients suffered from postoperative nausea and vomiting will be recorded in each group. | 24 hours postoperative

SECONDARY OUTCOMES:
antiemetic consumption | 24 hours postoperatively
  frequency of antiemetic consumption will be determined

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Haney Baumey, Banhā
  - Neveen Kohaf, Tanta

IPD SHARING:
Plan to Share IPD: Yes
data could be shared upon reasonable request from principal investigator
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Bauiomy H, Kohaf NA, Saad M, Rashed ZF, Abosakaya AM. Study the Effect of Intraperitoneal Dexamethasone, Dexmedetomidine, and Their Combination on PONV After Laparoscopic Cholecystectomy: A Randomized Triple-Blind Trial. Anesthesiol Res Pract. 2025 Feb 24;2025:4976637. doi: 10.1155/anrp/4976637. eCollection 2025. PMID 40041104